CLINICAL TRIAL: NCT02406612
Title: X-Seal 6F Vascular Closure Device EU Post-Market Clinical Follow-Up Protocol
Brief Title: X-Seal EU Post-Market Clinical Follow-Up Protocol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Essential Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: PSD-028
Record Dates: First submitted 2015-03-24; First posted 2015-04-02 (Estimated); Results first posted 2018-10-29 (Actual); Last update posted 2018-10-29 (Actual); Status verified 2018-01

CONDITIONS: Femoral Arteriotomy Closure
Keywords: Vascular Closure Device; Femoral Artery Closure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- X-Seal 6F Vascular Closure Device (Experimental): The X-Seal 6F Vascular Closure device will be used to achieve hemostasis in both diagnostic and interventional procedures using up to a 6F procedure sheath.
  Interventions: Device: X-Seal 6F Vascular Closure Device

INTERVENTIONS:
Device: X-Seal 6F Vascular Closure Device

SUMMARY:
The study is designed to prospectively collect data on and confirm the safety and effectiveness of the X-Seal 6F Vascular Closure System in reducing time to hemostasis and time to ambulation for patients who have undergone diagnostic or interventional catheterization procedures using up to 6F sheaths when compared with standard compression techniques using data from literature surveys.

ELIGIBILITY:
Inclusion Criteria:

* Candidate for non-emergent diagnostic or interventional cardiac catheterization via a femoral sheath ≤6F.
* Age ≥18 years.
* Understand and sign the study specific written informed consent form.
* In the investigator's opinion, the patient is suitable for the X-Seal vascular closure device, conventional hemostasis techniques and participation in an investigational trial.
* Eligible for sheath removal in the catheterization lab.

Exclusion Criteria:

* Patients who are known to be pregnant or lactating.
* Patients who are immunocompromised.
* Prior target artery closure with any vascular closure device or closure with manual compression win 30 days prior to this procedure.
* Patients with significant anemia (hemoglobin <10 g/DL, Hct<30).
* Patients who are morbidly obese or cachectic (BMI >40 or <20 kg/m2).
* Patients with Systolic Blood Pressure >180 mmHg, unless Systolic Pressure can be lowered by pharmacological agents prior to closure
* Patients who are currently participating in another clinical trial of an investigational drug or device that has not concluded the follow-up period.
* Patients with a baseline INR > 1.5 (e.g. coumadin therapy).
* Patients with a known bleeding disorder including thrombocytopenia (platelet count <100,000 cells/UL), thrombasthenia, hemophilia, or von Willebrand's disease.
* Patients with small femoral arteries (<4 mm), femoral artery stenosis resulting in a vessel diameter <4 mm, or patients with severe peripheral vascular disease.
* Patients with puncture site believed to be in the profunda femoris, superficial femoral artery, or at the bifurcation of the arteries.
* Common femoral artery with fluoroscopically visible calcium.
* Femoral arteries that are suspected to have experienced a back wall puncture or that underwent >one (1) arterial puncture during the catheterization procedure.
* Patients having a complication(s) at the femoral artery access site pre-sheath removal including hematoma, pseudoaneurysm, or arterio-venous fistula.
* Patients in whom continued heparin or other anticoagulant/antiplatelet therapy is planned (with the exception of Glycoprotein IIb/IIIa receptor blockers) following completion of the catheterization procedure.
* Patients whose ACT is >300 seconds prior to removal of the guiding catheter.
* Patients who cannot adhere to or complete the investigational protocol for any reason including but not limited to geographical residence or life threatening disease.
* Prior femoral vascular surgery or vascular graft in region of access site.
* Patient is unable to ambulate at baseline.
* Acute ST-elevation MI within 48 hours prior to procedure.
* Active systemic or cutaneous infection or inflammation
* Patients with unilateral or bilateral lower extremity amputation
* Patients with renal insufficiency (serum creatinine >2.5 mg/dl)
* Patients with marked tortuosity of the femoral or iliac artery
* Patients in whom bacterial contamination of the procedure sheath or surrounding tissues may have occurred as this may result in infection
* Patients in whom the puncture site is located above the most inferior border of the epigastric artery (IEA) and/or above the inguinal ligament based upon bony landmarks, since such a puncture site may result in a retroperitoneal hematoma/bleed. Perform a femoral angiogram to verify the location of the puncture site
* Patients with known allergies to beef products, collagen and/or collagen products, or polyglycolic or polylactic acid polymers
* Patients with known allergy to stainless steel or nickel. See MRI information in the IFU.
* Patients undergoing therapeutic thrombolysis
* Patients punctured through a vascular graft

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2015-04; Primary Completion 2016-02 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - University of Lubeck Hospital, Lübeck
  - University of Rostock Hosptial, Rostock

RESULTS

PARTICIPANT FLOW:
Groups:
- Diagnostic: Patients treated with X-Seal device that were undergoing a diagnostic catheter procedure.
- Interventional: Patients treated with X-Seal device that underwent an interventional catheter procedure.
Period: Overall Study
Arm/Group | Diagnostic | Interventional
Started | 26 | 21
Completed | 22 | 17
Not Completed | 4 | 4
Not completed — Screening Failure | 3 | 0
Not completed — Intra-procedural Exclusion | 1 | 3
Not completed — Guidewire Failure | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Diagnostic | Interventional | Total
Number analyzed (Participants) | 22 | 17 | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.1 (13) | 66.3 (11.8) | 65.1 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 4 | 12
  Male | 14 | 13 | 27
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 22 | 17 | 39
Ankle-Brachial Index (ABI) [Mean (Standard Deviation); unit: Ratio] | 1.1 (0.1) | 1.0 (0.2) | 1.0 (0.1)

OUTCOME MEASURES:

1. Primary Outcome: Major Complications
Description: The rate of major complications within approximately 30 days following the procedure.
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Groups:
- Diagnostic: Patients treated with X-Seal device that were underwent a diagnostic catheter procedure.
Arm/Group | Diagnostic | Interventional
Number analyzed (Participants) | 23 | 18
Participants | 0 | 0

2. Primary Outcome: Time-to-Hemostasis
Description: Time to hemostasis will be measured as the time from removal of the guiding catheter to the time of cessation of common femoral artery bleeding.
Time Frame: Time to hemostasis will be measured as the time from removal of the guiding catheter to the time of cessation of common femoral artery bleeding, assessed up to 2 hours.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Diagnostic | Interventional
Number analyzed (Participants) | 22 | 17
Minutes | 0.36 (1.14) | 0.65 (1.37)

3. Secondary Outcome: Time-to-Ambulation
Description: The time from end of the procedure until the patient ambulates for the first time.
Time Frame: Ambulation will be assessed 1.5 hours after removal of the access sheath for Diagnostic Patients, and 3 hours after procedure sheath removal for Interventional Patients.
Population: Subjects for whom ambulation data are available
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Diagnostic | Interventional
Number analyzed (Participants) | 20 | 16
hours | 3.52 (1.09) | 3.16 (1.14)

4. Secondary Outcome: Adverse Events
Description: The rate of adverse events within approximately 30 days following the procedure. All AEs counted, whether or not device-related.
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Diagnostic | Interventional
Number analyzed (Participants) | 26 | 21
Participants | 2 | 8

ADVERSE EVENTS:
Time Frame: 30 days post-procedure
Groups:
- Diagnostic: Patients treated with X-Seal device that underwent a diagnostic catheter procedure.
Arm/Group | Diagnostic | Interventional
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/21
Serious Adverse Events (participants affected / at risk) | 1/26 | 4/21
Other Adverse Events (participants affected / at risk) | 1/26 | 6/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Diagnostic (N=26) | Interventional (N=21)
New catheterization (Cardiac disorders) | 0 | 1
Hypertension (Cardiac disorders) | 0 | 1
Pancreatitis (Endocrine disorders) | 1 | 0
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Arrhythmia (Cardiac disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Diagnostic (N=26) | Interventional (N=21)
Hematoma (Vascular disorders) | 0 | 3
Pressure at access site (Vascular disorders) | 1 | 1
Guidewire tip detachment (Product Issues) | 0 | 1
Bleeding from contralateral access site (Vascular disorders) | 0 | 1
Pain at access site (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No